CLINICAL TRIAL: NCT04474054
Title: FARA-Free: A Single Arm Pilot Study of Pulsed Field Ablation in the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: A Single Arm Pilot Study of Pulsed Field Ablation in the Treatment of Paroxysmal Atrial Fibrillation
Acronym: FARA-Free
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0766
Record Dates: First submitted 2020-07-07; First posted 2020-07-16 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Catheter Ablation; Paroxysmal Atrial Fibrillaltion; Pulmonary Vein Isolation; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- FARAPULSE Ablation System Plus (Experimental): Ablation using the FARAPULSE Ablation System Plus
  Interventions: Device: Catheter ablation to treat paroxysmal atrial fibrillation

INTERVENTIONS:
Device: Catheter ablation to treat paroxysmal atrial fibrillation — A pulmonary vein isolation will be performed using catheter ablation

SUMMARY:
The objective of this pilot study is to confirm that endocardial ablation using the FARAPULSE Ablation System Plus with commercial design devices is both safe and effective for treating drug-resistant paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm safety and effectiveness pilot study. Subjects will undergo percutaneous PFA ablation for pulmonary vein isolation and at the clinical discretion of the investigator receive PFA ablation of additional arrhythmogenic locations. Subjects will be followed at 7 days (telephonic), 30 days, 90 days, 6 months and 12 months for adverse events, recurrence of arrhythmia after a 90-day Blanking Period and other relevant outcome measures.

ELIGIBILITY:
Inclusion Criteria:Study subjects are required to meet all the following inclusion criteria to participate in this study:

1. Patients with documented drug resistant symptomatic PAF
2. Patients who are ≥ 18 and ≤ 75 years of age on the day of enrollment.
3. Patient participation requirements:

   1. Lives locally.
   2. Is willing and capable of providing Informed Consent to undergo study procedures.
   3. Is willing to participate in all examinations and follow-up visits and tests associated with this clinical study.

Exclusion Criteria: Subjects will be excluded from participating in this study if they meet any one of the following exclusion criteria:

1. AF that is:

   1. Persistent
   2. Secondary to electrolyte imbalance, thyroid disease, alcohol abuse or other reversible / non-cardiac causes
   3. Longstanding
2. Left atrial anteroposterior diameter ≥ 5.0 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT)
3. Any of the following cardiac procedures, implants or conditions:

   1. Clinically significant arrhythmias other than AF, AFL or AT
   2. Previous endocardial or epicardial ablation or surgery for AF
   3. Hemodynamically significant valvular disease
   4. Prosthetic heart valve
   5. Heart Failure for example NYHA Class III or IV CHF, LVEF <40%, Heart failure hospitalization
   6. Atrial or ventricular septal defect closure
   7. Atrial myxoma
   8. Left atrial thrombus
   9. Left atrial appendage device or occlusion
   10. Pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices
   11. Significant or symptomatic hypotension
   12. Bradycardia or chronotropic incompetence
   13. History of pericarditis
   14. History of rheumatic fever
   15. History of congenital heart disease with any residual anatomic or conduction abnormality
   16. Any pulmonary vein abnormality, stenosis or stenting
4. Any of the following cardiovascular procedures, implants, or conditions:

   a. Within the 3 months preceding enrollment:

   i. Myocardial infarction

   ii. Unstable angina

   iii. Percutaneous coronary intervention

   iv. Treatment with amiodarone

   b. Within the 6 months preceding enrollment:

   i. Heart surgery

   ii. Stroke or TIA

   iii. Any thromboembolic event

   iv. Carotid stenting or endarterectomy

   v. Pericarditis or pericardial effusion

   c. Within the 12 months following enrollment:

   i. Any likelihood of cardiac surgery or transplant
5. History of blood clotting or bleeding abnormalities.
6. Contraindication to, or unwillingness to use, systemic anticoagulation
7. Contraindications to both CT and MRI
8. Sensitivity to contrast media not controlled by premedication
9. Women of childbearing potential who are pregnant, lactating, not using birth control or planning to become pregnant during the anticipated study period
10. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or confound data or its interpretation, including but not limited to

    1. Body mass index (BMI) > 40
    2. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
    3. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or significant dyspnea
    4. Renal insufficiency with an estimated creatinine clearance < 30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
    5. Active malignancy or history of treated cancer within 24 months of enrollment
    6. Clinically significant gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
    7. Clinically significant infection
    8. Predicted life expectancy less than one year
11. Clinically significant psychological condition that in the investigator's opinion would prohibit the subject's ability to meet the protocol requirements
12. Current or anticipated enrollment in any other clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ante Anic, Principal Investigator — University Hospital of Split
Locations (1):
- KBC Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intent To Treat (ITT): Enrolled subjects who undergo one or more ablation at the index procedure using the study device.
Period: Overall Study
Arm/Group | Intent To Treat (ITT)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intent To Treat (ITT)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Croatia | 15
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.3 (3.8)
Time Between First Documented Atrial Fibrillation Diagnosis and Enrollment [Mean (Standard Deviation); unit: months] — Population: Data unavailable for all 10 subjects
  months
    number analyzed (Participants) | 5
    (all) | 12.2 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Occurence of Device-or Procedure-related Early and Late-onset of Serious Adverse Events
Description: Includes serious adverse events which are device- or procedure-related, and as define din Composite Safety Endpoint definition table occurring within 7 days of the index procedure or hospital discharge, whichever is later, and diagnosed at any time during the follow-up period.
Time Frame: 7 days to12 Months
Measure: Count of Participants; unit: Participants
Groups:
- FARAPULSE Endocardial Ablation: Subjects who are treated with the FARAPULSE Endocardial Ablation System for paroxysmal atrial fibrillation.
  FARAPULSE Endocardial Ablation System: Endocardial ablation using the FARAPULSE Endocardial Ablation System.
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 15
Participants | 0

2. Primary Outcome: Freedom From Recurrence of Symptomatic Atrial Fibrillation, Atrial Tachycardia or Atrial Flutter
Description: Includes both acute procedural success (successful electrical isolation of set of lesions around the ostia of all pulmonary veins) and therapeutic success (Re-treatment for AF with ablation using study devices, or if necessary, a commercially approved ablation device after a 3 month blanking period constitute a treatment failure.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Endocardial Ablation
Number analyzed (Participants) | 15
Participants | 10

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | FARAPULSE Endocardial Ablation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Endocardial Ablation (N=15)
Atrial Tachycardia (Cardiac disorders) | 2 (2)
Supraventricular Tachycardia (Cardiac disorders) | 2 (2)
Transient Ischemic Attack (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Endocardial Ablation (N=15)
Hospitalization (Surgical and medical procedures) | 4 (4)
Corona Virus Infection (Infections and infestations) | 2 (2)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Vascular Access Complication (General disorders) | 4 (4)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT04474054/Prot_SAP_000.pdf